CLINICAL TRIAL: NCT01634698
Title: Responsiveness of RDR Test to Assess Hepatic Vitamin A Stores in Chronic Liver Disease
Brief Title: Relative-dose-response Test (RDR) Adaptation for Chronic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Gabriela Villaca Chaves, PhD, PhD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CEPHUCFF 06801
Record Dates: First submitted 2012-06-25; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Liver Disease
Keywords: chronic liver disease; cirrhosis; vitamin A; RDR test; retinol-binding protein
MeSH Terms: conditions — Fibrosis | interventions — retinol palmitate; United Nations; Vitamin A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RDR test (1500 UI vitamin A) (Experimental): 81 patients with several etiologies of liver cirrhosis at different stages in the progression of the disease received 1500 UI retinyl palmitate dosage at T0 (blood sample taken following a 12-hour fast). Following supplementation, we took further blood samples five and seven hours later (T5 and T7).
  Interventions: Dietary Supplement: retinyl palmitate (UNICEF, Melbourne, Australia)
- RDR test (2500 IU vitamin A) (Experimental): 81 patients with several etiologies of liver cirrhosis at different stages in the progression of the disease received 2500 UI retinyl palmitate dosage at T0 (blood sample taken following a 12-hour fast). Following supplementation, we took further blood samples five and seven hours later (T5 and T7).
  Interventions: Dietary Supplement: retinyl palmitate (UNICEF, Melbourne, Australia)

INTERVENTIONS:
Dietary Supplement: retinyl palmitate (UNICEF, Melbourne, Australia) — the patients received an oral dose of 1500 IU or 2500 IU, once.
  Other Names: vitamin A

SUMMARY:
The relative-dose-response test (RDR) is considered to be the most accurate method for evaluating vitamin A nutritional status (VANS) in patients suffering from liver disease, as it infers the reserves of the vitamin in the liver. However, for the RDR test to reflect VANS in patients suffering from chronic liver disease, factors inherent to the disease need to be considered, such as possible malabsorption, advanced age, a drop in synthesis and/or the release of retinol binding protein (RBP), which would result in an inadequate response to the RDR test. Thus, the objective of present study is to assess the adequacy of two different protocol for using the RDR test in patients with cirrhosis and cirrhosis-related hepatocellular carcinoma.

Methods: The sample group was comprised of 178 patients at Federal University of Rio de Janeiro University Hospital (111 men) with several etiologies of liver cirrhosis at different stages in the progression of the disease. They were sorted into two groups, according to the retinyl palmitate dosage (1500 IU or 2500 IU) received at T0 (blood sample taken following a 12-hour fast). Following supplementation, the investigators took further blood samples five and seven hours later (T5 and T7). The investigators assessed VANS via concentrations of serum retinol and RBP, as well as by way of the RDR test. The cutoff points the investigators used for denoting inadequacy in the indicators retinol and RDR were, respectively, < 1.05 µmol/L and ≥ 20%. To classify the degrees of severity of the disease the investigators used the criteria established by Child & Pugh (1973).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of liver cirrhosis of viral etiology, alcoholic or metabolic action

Exclusion Criteria:

* malabsorption syndromes
* moderate or severe infection
* diabetes mellitus using insulin renal, cardiac or respiratory
* therapeutic doses of vitamin A in the 6 months prior to data collection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in retinol status (RDR test) at 5 and/or 7 hour after supplementation | RDR will be calculated for the two intervention groups (1500 or 2500 IU vitamin A), for the two moments of blood sampling, 5 and 7 hours after supplementation.
  Therapeutic response is evaluated by means of circulating serum retinol, 5 and 7 hours after the administration of vitamin A. The RDR was calculated by the following formula, using the values of serum retinol in the three times of blood collection (Loerch et al., 1979), expressed in percentages:
  RDR (%) = [(A0-Ax) / Ax] x100 where A0 is the serum retinol at time 0 (fasting) and Ax is the serum retinol 5 or 7 h after administration of vitamin A. It was used as the RDR cutoff ≥ 20%, indicating indirect hepatic reserve inadequate

SECONDARY OUTCOMES:
serum retinol-binding protein (RBP) | RBP were analyzed at baseline, 5 and 7 hours after supplementation as a variable that explain the appropriate response or failure to respond to the RDR test.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela V Chaves, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Gabriela Villaça Chaves, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Peres WA, Chaves GV, Goncalves JC, Ramalho A, Coelho HS. Vitamin A deficiency in patients with hepatitis C virus-related chronic liver disease. Br J Nutr. 2011 Dec;106(11):1724-31. doi: 10.1017/S0007114511002145. Epub 2011 Jun 8. PMID 21736776